CLINICAL TRIAL: NCT06689098
Title: Diagnostic Accuracy of Magnetocardiography in Inflammatory Cardiomyopathies: A Comparison With Noninvasive Cardiovascular Magnetic Resonance (CMR) and Invasive Endomyocardial Biopsy
Brief Title: Magnetocardiography as a Diagnostic Screening Tool for Myocarditis and Other Types of Cardiomyopathy
Acronym: MagMa
Status: Completed | Type: Observational
Sponsor: German Heart Institute (Other)
Collaborators: Berlin Institute of Health at Charité (Unknown); Charite University, Berlin, Germany (Other); Biomagnetik Park Holding GmbH (Unknown)
Responsible Party: Principal Investigator, Bettina Heidecker, Head of Heart Failure and Cardiomyopathy, German Heart Institute
Other Study IDs: Magma-Study
Record Dates: First submitted 2024-10-23; First posted 2024-11-14 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Cardiomyopathies
Keywords: Magnetocardiography; Myocarditis; Inflammatory Cardiomyopathy; Cardiomyopathy; Biomarker; Heart Failure; Invasive diagnostic procedure; Noninvasive, endomyocardial biopsy; cardiac magnetic resonance imaging
MeSH Terms: conditions — Cardiomyopathies; Myocarditis; Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with suspected inflammatory cardiomyopathy: Adult patients experiencing cardiac symptoms such as chest pain or pressure, dyspnea on exertion, and heart racing are included after rule out of obstructive coronary artery disease by coronary angiography (ANOCA). Patients have to be stable enough to undergo advanced imaging and magnetocardiography measurements. Patients on immunosuppressive therapy and/or with intracardiac metal devices are excluded.
  110 patients for this group are planned.
  Interventions: Diagnostic Test: Magnetocardiography scan
- Cardiac Healthy Controls: Healthy individuals with no history of cardiac disease and unremarkable physical exam, 12-lead ECG, and echocardiography.
  220 patients for this group are planned

INTERVENTIONS:
Diagnostic Test: Magnetocardiography scan — The MCG system utilizes an array of 64 highly sensitive magnetic sensors known as superconducting quantum interference devices (SQUIDs). These sensors are placed in a shielded environment to reduce interference from external electromagnetic sources. SQUIDs capture variations in the heart's magnetic field throughout the cardiac cycle and correlate these changes with the QRS complex. To filter out electromagnetic noise, several frequency filters are applied. The measurements provide a three-dimensional view of the magnetic field, which is used to generate a composite vector representing the primary electrical axis of the heart. In assessing inflammatory cardiomyopathies, the focus is on the vector associated with the T-wave of the action potential, i.e. the vector from the T-wave beginning to the maximum (T-beg-Tmax interval). A T-wave/MCG vector T-beg-Tmax value ≥ 0.051 has been identified as indicative of pathology, as demonstrated in our previous research.
  Groups: Patients with suspected inflammatory cardiomyopathy

SUMMARY:
Accurate and rapid screening is an unmet medical need to address the increasing demand for advanced diagnostic workup in patients with suspected cardiomyopathy. Due to an overwhelmed health care system, advanced imaging is not always immediately available leading to underdiagnosis and progression of cardiomyopathies to advanced stages and sudden death. The investigator's recently demonstrated in a retrospective study that magnetocardiography (MCG) could be a suitable tool to detect inflammatory and other types of cardiomyopathies in a highly effective manner and without any safety issues. In this study, the investigator's test diagnostic accuracy of MCG prospectively.

DETAILED DESCRIPTION:
Inflammatory cardiomyopathy is one of the most common causes of sudden cardiac death in young adults, as it frequently remains undetected. Also, it is a common cause of heart failure, which may lead to circulatory collapse, requiring mechanical circulatory support or heart transplant. Some patients may require immunosuppression in addition to standard heart failure therapy. Early initiation of therapy is crucial for optimal outcomes.

Inflammatory disease of the heart muscle/inflammatory cardiomyopathy can be challenging to diagnose because it often requires expensive, time intense, and sometimes invasive testing, such as cardiac magnetic resonance imaging (MRI) and endomyocardial biopsies (EMB). As a result, there is an unmet clinical need for low threshold diagnostic screening in patients with suspected cardiomyopathy.

In this study the investigator's evaluate the diagnostic accuracy of magnetocardiography (MCG) in detecting inflammatory and other types of cardiomyopathy. Diagnostic accuracy will be compared to results from advanced imaging (cardiac magnetic resonance (CMR) imaging and/or positron emission computed tomography (PET-CT)) and where available to histology from endomyocardial biopsy/EMB.

CMR provides comprehensive structural and functional data while detecting consequences of inflammation, such as edema and late gadolinium enhancement. PET-CT detects the level of activity and the extent of inflammation through measurement of glucose metabolism. However, it cannot be applied frequently because of the associated radiation exposure. EMB is the gold standard for definitive diagnosis of inflammatory cardiomyopathy and is crucial for initiation of immunosuppressive therapy, as active viral infection should be excluded. However, the limited diagnostic yield due to sampling error and risk of potential complications limit its use to selected cases where there is a high suspicion that specific treatment may be necessary.

MCG is based on detecting the movement of ions in the myocardium. When an action potential in the heart is generated, it creates voltage changes and consequently an electromagnetic field. The strength and direction of this field are affected by the flow of ions both inside and outside the cells. Typically, the magnetic field produced by the heart ranges from from 10-15 to 11-11 Tesla.

MCG uses a superconducting quantum interference device (SQUID) to detect the electromagnetic field of the heart (up to 10*-15 Tesla). Measurements take place during the ascending T wave of the cardiac cycle. A vector score > 0.051 was determined to be pathologic in our recently published retrospective study. The investigator's will assesss diagnostic accuracy of MCG relative to cardiac magnetic resonance imaging (CMR) or positron emission computed tomography (PET-CT) and endomyocardial biopsy (EMB). Results from EMB take precedence over advanced imaging. Results from MCG will be independently assessed by two trained professionals blinded to the clinical diagnosis, with a third expert to adjudicate in cases of disagreement.

The MCG system utilizes an array of 64 highly sensitive magnetic sensors known as superconducting quantum interference devices (SQUIDs). These sensors are placed in a shielded environment to reduce interference from external electromagnetic sources. SQUIDs capture variations in the heart's magnetic field throughout the cardiac cycle and correlate these changes with the ECG. To filter out electromagnetic noise, several frequency filters are applied. The measurements provide a three-dimensional view of the magnetic field, which is used to generate a composite vector representing the primary electrical axis of the heart. In assessing inflammatory cardiomyopathies, the focus is on the vector associated with the T-wave of the action potential, specifically between the beginning of the T-wave on a 12-lead ECG to the maximum of the T-wave (T-beg-Tmax interval). A T-wave/MCG vector T-beg-Tmax value ≥ 0.051 has been identified as indicative of pathology, as demonstrated in our previous research (Brala et al, JAHA, 2023, PMID: 36744683).

The goal of this project is to validate the diagnostic accuracy of MCG for diagnosing inflammatory and other types of cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with angina-like symptoms after exclusion of coronary artery disease

Exclusion Criteria:

* Presence of intracardiac metal devices and prior treatment with immunosuppressants

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The healthy controls do not have any history of cardiac disease. Standard examiniations ensure that there are no undiagnosed conditions.
Sampling Method: Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Accurate diagnosis of inflammatory cardiomyopathy | MCG is obtained at the time of clinical presentation. Accuracy of diagnosis by MCG is tested with the current diagnostic gold standard methods: CMR, PET-CT and/or EMB, when clinically indicated.
  The main outcome is the correct diagnosis of an inflammatory cardiomyopathy, the noninvasive gold standard cardiac magnetic resonance imaging or invasive gold standard endomyocardial biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Heidecker, MD, Principal Investigator — Deutsches Herzzentrum der Charité
Locations (1):
- Deutsches Herzzentrum der Charité, Steglitz, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Data from the study can be made available upon request from the principal investigator PD Dr. med. Bettina Heidecker in a de-identified form. A data use agreement must be signed before access to data. Access is only granted to academic staff.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: see above
Access Criteria: see above